CLINICAL TRIAL: NCT00355576
Title: Phase II Combination Therapy Selection Trial in Amyotrophic Lateral Sclerosis
Brief Title: Combination Therapy Selection Trial in Amyotrophic Lateral Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: ALS Association (Other); Pfizer (Industry)
Responsible Party: Paul H. Gordon, Columbia University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAAB6334; ALSA ID#920 (Other: CUMC)
Record Dates: First submitted 2006-07-21; First posted 2006-07-24 (Estimated); Last update posted 2011-02-01 (Estimated); Status verified 2011-01

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; Celecoxib; Creatine; Minocycline; Combination; Selection; ALS; Motor Neuron Disease
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; cyclopia sequence; Motor Neuron Disease | interventions — Celecoxib; Creatine; Minocycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Minocycline + Creatine (Experimental): Minocycline 100 mg BID and Creatine 10 g BID
  Interventions: Drug: Creatine; Drug: Minocycline
- Celecoxib + Creatine (Experimental): Celecoxib 400 mg BID and Creatine 10 g BID
  Interventions: Drug: Celecoxib; Drug: Creatine

INTERVENTIONS:
Drug: Celecoxib — Celecoxib 400 mg BID with creatine 10 g BID if randomized to the Celecoxib + Creatine study arm.
  Arms: Celecoxib + Creatine
Drug: Creatine — 10 g BID for either study arm
Drug: Minocycline — Minocycline 100 mg BID with creatine 10 g BID if randomized to the Minocycline + Creatine study arm
  Arms: Minocycline + Creatine

SUMMARY:
The objective of this study is to compare two combinations of drugs, minocycline and creatine or celecoxib and creatine, in a phase II trial designed to determine which combination is more effective for ALS.

DETAILED DESCRIPTION:
Excess free radicals, energy mishandling, excitotoxicity, activation of cell death pathways and inflammation likely all contribute to neurodegeneration in ALS. Past trials may have been negative in part because they tested single agents, usually influencing only one mechanism of cell death. Combinations of agents that affect different and multiple mechanisms of neurodegeneration may be necessary to reach meaningful outcomes in trials of ALS.

This trial has several unique features. First, it compares the neuroprotective potential of two combinations of agents that impact multiple mechanisms of cell death. The combinations of minocycline/creatine and celecoxib/creatine are the only agents that have had additive effects in the mouse model of ALS, reducing neurodegeneration and prolonging survival more than individual agents alone. Second, it uses an important new phase II selection trial design to determine which combination is superior. Not only does this trial test combination therapy, but there is no placebo, so everyone who enrolls in the trial will receive active treatment.

Minocycline, creatine and celecoxib have been tested individually and have been shown to be safe in patients with ALS. This will be the first time human trials will be conducted with combinations of minocycline/creatine and celecoxib/creatine.

We will compare combinations of drugs in a phase II trial design to determine which combination is superior. If successful, this trial will lead directly to a phase III trial of the selected combination. If the design is found useful, this trial will lead to larger phase II selection trials assessing greater numbers of agents simultaneously, thereby improving the efficiency of drug screening in ALS.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of possible, laboratory-supported probable, probable or definite ALS, according to modified EL Escorial criteria
* FVC greater or equal to 60% at the screening visit
* Symptom onset within 5 years
* 21 to 85 years of age
* If patients are taking riluzole, they must be on a stable dose for at least the past thirty days
* A woman of childbearing age, must be nonlactating and surgically sterile or using an effective method of birth control (barrier method) and have a negative pregnancy test
* Able to maintain adequate hydration levels defined as 6-8 cups (8ounces/cup) of water or a non-caffeinated beverage per day
* Willing and able to give signed informed consent that has been approved by an Institutional Review Board (IRB)

Exclusion Criteria:

* Tracheotomy and mechanical ventilation
* Diagnosis of other neurodegenerative diseases (Parkinson's disease, Alzheimer's disease, etc)
* Unstable medical illness (coronary artery disease, advanced cancer, active esophageal or gastroduodenal ulcers, etc) in the last one year
* Systemic Lupus Erythematosis
* FVC < 60%
* Pregnancy or lactation
* Allergy to minocycline, tetracyclines, celecoxib, sulfonamides, NSAIDS, or creatine
* History of congestive heart failure
* Renal disease [baseline Cr > 1.5 (men) or 1.2 (women)]
* History of significant hepatic disease (baseline AST/ALT or bilirubin > 1.5x normal)
* Use of an investigational agent within thirty days of enrollment
* First degree relative with ALS or gene identified familial ALS
* Inability or unwillingness to maintain adequate daily hydration (defined above)
* Limited mental capacity such that the patient cannot provide written informed consent or comply with evaluation procedures.
* History of recent alcohol or drug abuse or noncompliance with treatment or other experimental protocols.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2006-07; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
ALS Functional Rating Scale Revised (ALSFRS-R) completed monthly during trial. | Up to 6 months from the start of treatment

SECONDARY OUTCOMES:
Forced Vital Capacity, Quality of Life, Timed Get Up and Go performed monthly. Survival and measures of safety throughout the trial. | Up to 6 months from the start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Paul H Gordon, MD, Principal Investigator — Columbia University
Locations (19):
- United States (19):
  - Phoenix Neurological Associates, Phoenix, Arizona
  - UCLA, Los Angeles, California
  - University of California Irvine, Orange, California
  - California Pacific Medical Center, San Francisco, California
  - Mayo Clinic Florida, Jacksonville, Florida
  - Medical College of Georgia, Augusta, Georgia
  - University of Illinois, Chicago, Illinois
  - University of Kansas, Kansas City, Kansas
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - UMDNJ, New Brunswick, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Beth Israel, New York, New York
  - Columbia University, New York, New York
  - Duke University, Durham, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Vermont, Burlington, Vermont

REFERENCES:
- [Background] Klivenyi P, Kiaei M, Gardian G, Calingasan NY, Beal MF. Additive neuroprotective effects of creatine and cyclooxygenase 2 inhibitors in a transgenic mouse model of amyotrophic lateral sclerosis. J Neurochem. 2004 Feb;88(3):576-82. doi: 10.1046/j.1471-4159.2003.02160.x. PMID 14720207
- [Background] Zhang W, Narayanan M, Friedlander RM. Additive neuroprotective effects of minocycline with creatine in a mouse model of ALS. Ann Neurol. 2003 Feb;53(2):267-70. doi: 10.1002/ana.10476. PMID 12557297
- [Background] Cheung YK, Gordon PH, Levin B. Selecting promising ALS therapies in clinical trials. Neurology. 2006 Nov 28;67(10):1748-51. doi: 10.1212/01.wnl.0000244464.73221.13. PMID 17130405
- See also: Eleanor and Lou Gehrig MDA/ALS Research Center at Columbia University website — http://www.columbiaals.org
- See also: ALS Association Website — http://www.alsa.org